CLINICAL TRIAL: NCT03496649
Title: Feasability Study on the Use of Botulinum Toxin A in Primary Adductor Tendinopathies Refractory to Medical Treatment
Brief Title: Pubalgia and Adductor Tendinopathies Refractory to Medical Treatment
Acronym: PETRA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2014/21
Record Dates: First submitted 2017-08-03; First posted 2018-04-12 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Groin Injury; Tendinopathy
Keywords: Primary Adductor tendinopathies; Pubalgia; Botulinum toxin type A
MeSH Terms: conditions — Tendinopathy | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dysport (Experimental): Dysport administration by intramuscular injection Each patient will receive one dose of Dysport at Visit 1.
  At least 2 of the 4 muscles below will be injected, depending on which muscles are affected:
  250 IU for the gracilis muscle 200 IU for the pectineus muscle 300 IU for the adductor longus muscle 200 IU for the adductor brevis muscle
  These injections will be uni or bilateral, it will depend on clinical diagnosis.
  If necessary, the 4 muscles will be injected with a maximum of 1500U Dysport. The total dose cannot exceed 1500 units.
  Interventions: Drug: Dysport 500 Unit Powder for Injection

INTERVENTIONS:
Drug: Dysport 500 Unit Powder for Injection — Dysport administered by intramuscular injection

SUMMARY:
Pubalgia is a pain syndrome located in the groin area. This syndrome is mainly described in young male athletes and typically affect the superficial muscles defining the boundaries of the femoral triangle, i.e. gracilis, pectineus, adductor brevis and especially adductor longus, and less commonly the deep muscles.

Clinically, the pain is located in the inner aspect of the thigh, where the tendons attach onto the pubic symphysis. It is usually unilateral, and sometimes associated with neuropathic pain suggestive of obturator nerve irritation.

There is no official recommendation or expert consensus on the management of pubalgia. However, a few protocols recommend a period of rest with Non-Inflammatory Anti-Steroidien Drugs (NSAIDs), icing and massages, as well as rehabilitation with passive stretching and muscle reinforcement.

The use of botulinum toxin type A could be an option in cases of treatment failure. However, a feasibility study must be performed beforehand, and if results are positive, a controlled study on a larger cohort could be conducted.

The major potential impact is a great effective pain relief for patients with neurological diseases.

DETAILED DESCRIPTION:
The incidence of pubalgia in the literature varies, with large series reporting an incidence close to 5-10%, representing 15 to 18% of all injuries.

Recurrences are also common, affecting 30 to 35% of cases.

Once other differential diagnoses (such as spondylarthropathy, colorectal cancer, kidney disease…) have been ruled out, athletic pubalgia is typically divided into three main categories based on the site of the injury:

* Abdominal wall, the most common form, representing 38 to 50% of all cases;
* Pubic symphysis due to osteoarthropathy of the pubic bone caused by repetitive stress injury, accounting for 10 to 15% of all cases of pubalgia;
* Adductor tendons, on which this study focuses, representing 22 to 38% of all cases of pubalgia, caused by repetitive tractions on the tendon insertions.

There is no official recommendation or expert consensus on the management of pubalgia. However, a few protocols recommend a period of rest with Non-Inflammatory Anti-Steroidien Drugs (NSAIDs), icing and massages, as well as rehabilitation with passive stretching and muscle reinforcement.

Neuromuscular reprogramming is then performed to stabilise the pelvis, followed by a progressive resumption of sporting activities, guided by the pain level.

Generally, 70 to 85% of patients are able to resume their sporting activities with this management protocol.

In 15 to 20% of cases of essential adductor tendinopathy, symptoms do not improve and the only currently validated solution is then a tenotomy, sometimes combined with partial tendon release in recurring cases.

Recent studies showed that the use of botulinum toxin type A (BTA) produces fairly positive results in chronic tendinopathies, such as epicondylitis. However, the efficacy of BTA injections in adductor tendinopathies has not been demonstrated consistently and a feasibility study must be conducted to address this question.

The hypothetical benefit of BTA in adductor tendinopathies is based on the toxin's known effects:

1. a purely analgesic effect, which reduces pain in the injected area within a few days. This type of chronic tendinopathy does not involve inflammation. The pain in such cases is most likely due to the action of neurotransmitters such as substance P and calcitonin gene-related peptide (CGRP). As BTA is known to inhibit the secretion of these neurotransmitters, this mechanism could explain the toxin's specific analgesic effect.
2. a muscle relaxant effect due to its action on the motor endplate, which reaches its maximum 6 weeks after the injection, and lasts 3 to 6 months.

The resulting muscle relaxation helps improve healing of the damaged tendon, and provides sustained analgesia.

A series including 39 cases showed that botulinum toxin is effective on hip adductor muscles following total hip arthroplasty, providing reduced muscle contracture and improved hip mobility without side effects.

The use of botulinum toxin type A could be an option in cases of treatment failure. However, a feasibility study must be performed beforehand, and if results are positive, a study on a larger cohort could be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 to 65 years old
* Patient with episode of adductor tendinopathy, refractory to appropriate medical treatment lasting 3 months
* Tendinopathy confirmed by clinical investigation, echography and MRI.
* Patient naïve to intramuscular botulinum toxin injections
* Patient able to self-evaluate pain on a VAS
* Intensity of exercise-induced pain > 5 on a VAS of 10
* Patient able to provide a signed informed consent freely for the study protocol and data collection

Exclusion Criteria:

* Subject participating or having participated in the last 3 months in another study which could interfere with the objective of the study
* Neuralgia
* Acute muscle injury
* Progressive disease at the time of inclusion
* Anticoagulant treatment: heparin administered with an electrical syringe or AVK therapy with effective doses

Exclusion criteria related to Dysport injection (botulinum toxin type A) :

* Known hypersensitivity to botulinum toxin type A or to any of the components in the formulation (20% human albumin solution, lactose monohydrate)
* Subject with a significant deficit of clinical or subclinical neuromuscular transmission (myasthenia or Lambert-Eaton syndrome)
* Treatment that directly or indirectly interferes with neuromuscular transmission (aminoglycosides, curare, anticholinesterase, aminoquinoline, cyclosporine, etc.)
* Previous surgery with curarisation less than a month ago
* History of neuromuscular disorders
* Pregnant or breastfeeding woman
* Women of child-bearing potential not using contraceptive methods during the study duration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-08-02 (Estimated); Study Completion 2020-08-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a pain reduction (VAS) | Between Day 80 and Day 90
  Proportion of patients with a pain reduction of over 50% compared to baseline, as shown by the average pain intensity measured between D80 and D90 on a Visual Analogic Scale (VAS) from 0 to 10 (0 = no pain; 10 = worst pain imaginable).
  Pain intensity will be daily collected by the patient in his patient's diary.

SECONDARY OUTCOMES:
Exercise-induced pain intensity (VAS) | Daily between Day 0 and Day 90
  Average intensity of exercise-induced pain evaluated daily by the patient on a VAS type numerical scale
Pain relief | On Day 30 and Day 90
  Percentage of patients with over 50% pain relief compared to baseline
Goal Attainment Scaling (GAS) | On Day 30 and Day 90
  Percentage of patients with over 50% GAS objective reached
Blazina clinical classification system | On Day 30 and Day 90
  Improvement of at least 1 point on the Blazina clinical classification system in 50% of patients
Adductor strength | On Day 30 and Day 90
  Preservation or improvement of adductor strength measured with a dynamometer and resumption of sport activity (Tegner activity level scale) in 50% of patients
Cure rate based on patients' self-evaluation | On Day 30 and Day 90
  Percentage of patients with over 50% cure rate based on the patients' self-evaluation of the improvement of their condition
Cure rate based on physician's evaluation | On Day 30 and Day 90
  Percentage of patients with over 50% cure rate based on the physicians' evaluation of the patients' improvement
Treatment | On Day 30 and Day 90
  Percentage of patients not asking for further treatment
Pain diary | On Day 30 and Day 90
  Determination of a break point on the pain intensity graph plotted by the physician, based on the pain diary completed by the patient.
HAGOS self-reported questionnaire | On Day 30 and Day 90
  Improvement on the 6 dimensions of the HAGOS self-reported questionnaire
Tolerance | Day 1, Day 7, Day 14, Day 30, Day 90
  Tolerance evaluation: description and frequency of adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided
Any exploitation of the data by Ipsen or for another research will be submitted to the preliminary agreement of CHU de Bordeaux and, in case of agreement, of a negotiated contract between the parties.